CLINICAL TRIAL: NCT07208448
Title: A Multi-Center, Prospective, First-In-Human Study to Evaluate the Initial Safety and Effectiveness of a Degradable Shoulder Spacer in Patients With Symptomatic Massive Rotator Cuff Tears
Brief Title: Voll Degradable Shoulder Spacer FIH Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Voll Medical Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 053CLD
Record Dates: First submitted 2025-09-18; First posted 2025-10-06 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Massive Rotator Cuff Tear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Voll Degradable Shoulder Spacer (Experimental)
  Interventions: Device: Voll Degradable Shoulder Spacer

INTERVENTIONS:
Device: Voll Degradable Shoulder Spacer — Voll Degradable Shoulder Spacer

SUMMARY:
The Voll Degradable Shoulder Spacer First-in-Human study aims to evaluate the initial safety, effectiveness, and clinical outcomes of a degradable shoulder spacer in over 50 years old patients with symptomatic massive rotator cuff tears (MRCT).

ELIGIBILITY:
Main Inclusion Criteria:

* Full thickness MRCT.
* Male or female patients ≥ fifty (50) years of age, in general good health, independent, and can comply with all post-operative evaluations and visits.

Main Exclusion Criteria:

* Documented evidence of a history of drug/alcohol abuse within 1 year of enrollment.
* Concurrent participation in any other investigational clinical study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Device-related Serious Adverse Events | Up to 12 months post-implantationץ
  Incidence of device-related serious adverse events (DRSAEs) related to the spacer.

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Assuta Ashdod Hospital, Ashdod
  - Ichilov (Sourasky Medical Center), Tel Aviv

IPD SHARING:
Plan to Share IPD: No